CLINICAL TRIAL: NCT03898076
Title: The Prediction of A1c Based on CGM Data Through Applying Machine Learning Approaches
Brief Title: Predictive A1c Based on CGM Data Using CGM Data
Acronym: A1c
Status: Completed | Type: Observational
Sponsor: Sidra Medicine (Other)
Responsible Party: Principal Investigator, Goran Petrovski, Goran Petrovski Clinical Professor, Sidra Medicine
Other Study IDs: 2019003271
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Flash Glucose Monitoring — Continuous Glucose Monitoring (CGM) values will be downloaded from CGM device for a period of 90 days.
Other: A1c — A1c levels will be collected from Hospital EMR prior to CGM data downoad
Other: Predictive A1c — Predictive A1c will be calculated based on the first 15 days of CGM data using time in range (TIR), coefficient of variation (CV), mean amplitude of glycemic excursion (MAGE), mean of daily differences (MODD), continuous overall net glycemic action (CONGA). Predictive A1c will be correlated with actual A1c.

SUMMARY:
Introduction. The hemoglobin A1C (HbA1c) reflects the average blood glucose level for last two to three months. Recent advancements in the sensor technology facilitate the daily monitoring of the blood glucose using CGM devices. The future prediction of the HbA1C based on the CGM data holds a critical significance in maintaining long term health of diabetes patients. A higher than normal value of the HbA1c greatly increases the likelihood of diabetes related cardiovascular disease.

Goal. The aim this study is to predict the HbA1c in advance by utilizing the CGM data through applying machine learning techniques. The outcomes of this research will assist in improving the health of diabetic patients.

Methods. This is a retrospective analysis. The investigators will de-identify and analyze 120 patients with T1D who using CGM sensor for last three months. Past 15 days of CGM data will be analyzed and different glucose variability features such as time in range (TIR), coefficient of variation (CV), mean amplitude of glycemic excursion (MAGE), mean of daily differences (MODD), continuous overall net glycemic action (CONGA) will be extracted. A machine learning model will calculate (predict) HbA1c in 2-3 months advance based on these 15 days of CGM data. To evaluate the performance of the proposed prediction model, predicted HbA1c will be compared with the real HbA1c.

DETAILED DESCRIPTION:
This is a retrospective analysis. The investigators will de-identify and analyze 120 patients with T1D using Continuous Glucose Monitoring (CGM) system for last three months. Past 15 days of CGM data will be analyzed and different glucose variability features such as time in range (TIR), coefficient of variation (CV), mean amplitude of glycemic excursion (MAGE), mean of daily differences (MODD), continuous overall net glycemic action (CONGA) will be extracted. A machine learning model will be developed to predict HbA1c in 2-3 months advance based on these 15 days of CGM data. The model is using linear regression, penalized regression (Ridge regression, Lasso regression and Elastic net regression) in combination gradient boosting to calculate predictive A1c

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Flash glucose Monitoring system

Exclusion Criteria:

* Less than 70% od CGM data in the last 90 days.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Type 1 Diabetes and Flash glucose monitoring
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The difference of Predictive A1c level from CGM data with Real A1c level from EMR | 3 months
  Difference (%) between Predicted A1c and laboratory A1c from the Electronic Medical Record

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Qaraqe, PhD, Principal Investigator — Hamad Bin Khalifa University, Doha; Hasan Abbas, PhD, Principal Investigator — TAMUQ, Doha
Locations (1):
- Sidra Medicine, Doha, Qa, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ball MJ, Lillis J. E-health: transforming the physician/patient relationship. Int J Med Inform. 2001 Apr;61(1):1-10. doi: 10.1016/s1386-5056(00)00130-1. PMID 11248599
- [Result] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Result] Ogurtsova K, da Rocha Fernandes JD, Huang Y, Linnenkamp U, Guariguata L, Cho NH, Cavan D, Shaw JE, Makaroff LE. IDF Diabetes Atlas: Global estimates for the prevalence of diabetes for 2015 and 2040. Diabetes Res Clin Pract. 2017 Jun;128:40-50. doi: 10.1016/j.diabres.2017.03.024. Epub 2017 Mar 31. PMID 28437734
- [Result] Rohlfing CL, Wiedmeyer HM, Little RR, England JD, Tennill A, Goldstein DE. Defining the relationship between plasma glucose and HbA(1c): analysis of glucose profiles and HbA(1c) in the Diabetes Control and Complications Trial. Diabetes Care. 2002 Feb;25(2):275-8. doi: 10.2337/diacare.25.2.275. PMID 11815495